CLINICAL TRIAL: NCT00002956
Title: A Phase I Pilot Trial to Evaluate the Toxicity of Allogeneic Epstein-Barr Virus Specific T-Lymphocytes for the Treatment of EBV-Associated Lymphoproliferative Diseases in Organ Transplant Recipients
Brief Title: Immunotherapy for Lymphoproliferative Diseases Associated With Epstein-Barr Virus in Patients Who Have Undergone Organ Transplants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065433; UAB-9739; IUMC-9611-37; NCI-V97-1176
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2012-11

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent childhood lymphoblastic lymphoma; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; T-cell large granular lymphocyte leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Recurrence; Leukemia, Large Granular Lymphocytic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- infusions of EBV specific cytotoxic T lymphocytes (Experimental): Donors undergo leukapheresis, and Epstein-Barr virus (EBV) specific cytoxic T lymphocytes are cultivated in vitro. Patients receive infusions of EBV specific cytotoxic T lymphocytes over 5 to 10 minutes on weeks 0, 2, and 4. Patients with stable disease and those achieving partial remission are followed weekly for signs of disease progression
  Interventions: Biological: allogeneic Epstein-Barr virus-specific cytotoxic T lymphocytes

INTERVENTIONS:
Biological: allogeneic Epstein-Barr virus-specific cytotoxic T lymphocytes

SUMMARY:
RATIONALE: Donor lymphocytes that have been exposed to Epstein-Barr virus may be able to help the body kill cancers associated with this virus.

PURPOSE: Phase I trial to study the effectiveness of Epstein-Barr virus-specific T cells derived from matched donors in organ transplant patients with lymphoproliferative diseases associated with Epstein-Barr virus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Examine the toxic effects of allogeneic Epstein-Barr virus (EBV) specific cytotoxic T lymphocytes (CTL) for the treatment of EBV lymphoproliferative diseases (LPD) in organ transplant recipients. II. Determine the level of in vivo expansion of allogeneic CTL and the period of time during which these CTL's can be detected in the blood of recipients of the T cell infusions.

OUTLINE: Donors undergo leukapheresis, and Epstein-Barr virus (EBV) specific cytoxic T lymphocytes are cultivated in vitro. Patients receive infusions of EBV specific cytotoxic T lymphocytes over 5 to 10 minutes on weeks 0, 2, and 4. Patients with stable disease and those achieving partial remission are followed weekly for signs of disease progression.

PROJECTED ACCRUAL: 10 patients will be accrued in this study.

ELIGIBILITY:
Inclusion criteria:

* Radiographic evidence of lymphadenopathy or lymphomatous lesions combined with clinical signs of Epstein-Barr virus lymphoproliferative disease (EBV LPD), such as fevers and lymphadenopathy
* following an organ transplant Persistent, progressive, or unresponsive disease despite decreased immunosuppression, chemotherapy, or radiation therapy EBV LPD must be of host origin
* At least 4 weeks
* Patients serologically hepatitis B and C positive may receive cytotoxic
* T- lymphocytes (CTL) from donors who are serologically positive for the same virus
* Must have an HLA identical or HLA haploidentical donor

Exclusion

* hepatic dysfunction SGOT/SGPT less than 2.5 times upper limit of normal (unless liver metastases present)
* Bilirubin less than 2.0 mg/dL
* renal dysfunction
* Creatinine clearance at greater than 50 mL/min
* cardiac dysfunction
* neurologic dysfunction
* pulmonary dysfunction
* patients developing EBV LPD who have a donor origin lymphoma
* HIV-1 positive
* Not capable of undergoing leukapheresis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1996-11; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Number of adverse events associated with administration of allogeneic Epstein-Barr virus (EBV) specific cytotoxic T lymphocytes (CTL) for the treatment of EBV lymphoproliferative diseases (LPD) in organ transplant recipients | baseline to x weeks post infusion
Mean length of time of allogeneic CTL during which these CTL's can be detected in the blood of recipients of the T cell infusions. | baseline to x weeks past infusion

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States